CLINICAL TRIAL: NCT00352872
Title: A Pilot Study of Cytochrome P450 Pharmacogenetics as a Predictor of Toxicity in Pre-Menopausal Women Receiving Doxorubicin and Cyclophosphamide in Early Breast Cancer
Brief Title: Pharmacogenetics as a Predictor of Toxicity in Pre-Menopausal Women Receiving Doxorubicin and Cyclophosphamide in Early Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: This study has been difficult to recruit.
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Bryan Schneider, Associate Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 0501-37
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: Pharmacogenetics; Toxicity; Pre-Menopausal; Women; Doxorubicin; Cyclophosphamide; Breast Cancer; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Plasma

SUMMARY:
The goal of this pilot study is to delineate the role of genetic variations in premature menopause, hot flashes, and other toxicities in a cohort of premenopausal women with early breast cancer.

Primary Objective- To ascertain the effect of common variant alleles of CYP450 2B6, 2C19, 2C9, and 3A5 in pre-menopausal women with breast cancer receiving anthracycline and cyclophosphamide based chemotherapy as it relates to occurrence of premature menopause (defined as more than 12 months of amenorrhea and serum estradiol and FSH levels consistent with post-menopausal status)

Secondary Objective #1- To obtain pilot data on the effect of common variant alleles of CYP450 2B6, 2C19, 2C9, and 3A5 in pre-menopausal women with breast cancer receiving anthracycline and cyclophosphamide based chemotherapy as it relates to occurrence of hot flash frequency, and other common toxicities of therapy requiring dose delay or reduction.

Secondary Objective #2- To obtain pilot data on the correlation of hot flashes with serum levels of serotonin, tryptophan, and their metabolites and with polymorphisms of the serotonin transporter and receptor genes.

DETAILED DESCRIPTION:
There is a clear survival benefit with the use of adjuvant cytotoxic therapy for most women with invasive breast cancer, even in those who have hormone receptor positive disease and receive adjuvant hormonal therapy with tamoxifen.1 In addition, several trials have shown a benefit for anthracycline based regimens over the more classic combination of cyclophosphamide, methotrexate, and 5-fluorouracil.1-4 The improved efficacy with taxanes in the adjuvant setting has more recently been demonstrated for patients with lymph-node positive disease.5-8 Despite clear survival benefits with cytotoxic therapy, the 10 year-disease specific mortality remains suboptimal at 69-78% and 49-53% for patients with and without lymph node involvement, respectively.9

Of the 180,000 women diagnosed with breast cancer in the United States, about one-fourth are pre-menopausal.10-13 Breast cancer clearly represents one of the most commonly diagnosed malignancies in this patient population. With the common use of adjuvant chemotherapy, long-term sequelae of treatment are becoming increasingly important. In addition to the acute toxicities of anthracycline and cyclophosphamide-based regimens,5 one side effect with both psycho-social and physical implications is pre-mature menopause.13-17 The frequency of menopause induced by poly-agent chemotherapy ranges from 34-89%.16,18,19 Multiple factors (both patient and drug-related) play a role in explaining this large variability. The age of the patient (at time of therapy),13,19,20 type of chemotherapy drugs,18,21 and duration and intensity22 of therapy all influence the overall likelihood of a patient prematurely entering menopause after therapy. In a previously reported study, age and systemic therapy were important variables in determining menopause in women with loco-regional breast cancer in multivariate analysis.19 Women with advancing age had a higher rate of menopause as expected. Hormonal therapy, and to a much greater degree, systemic therapy predicted early menopause. The combination of systemic and hormonal therapy appeared to have an additive effect on induction of menopause. Of importance, however, the added impact of hormonal therapy (when added to cytotoxic therapy) appears to play a minimal role in the induction of menopause when compared to cytotoxic therapy alone. It is also likely that intrinsic host genetic variability may also play a role as well. The variable ability to metabolize and clear a drug may, in part, affect efficacy and toxicity of these drugs and may ultimately impact the effect of the drug on ovarian function. One important example of this relates to polymorphisms in enzymes important in the clearance of the described drugs. To date, little work has been done to understand the importance of inter-individual, host specific variability on the risk of a breast cancer patient experiencing drug-induced, pre-mature menopause.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the breast and appropriate for treatment with Doxorubicin and Cyclophosphamide.
2. Age > 18 years and <45 years.
3. ECOG performance status of 0 to 2.
4. Signed informed consent.
5. Premenopausal: defined as regularly occurring menstrual cycles or serologic estradiol and FSH levels consistent with premenopausal status.

Exclusion Criteria:

1. Patients with distant metastatic disease will be excluded.
2. Pregnancy or breast feeding (women of childbearing potential must have a negative pregnancy test). Women of childbearing potential must be willing to consent to using effective contraception (oral contraceptive pill or implant or barrier method) while on treatment and for a 30 days after taking the last dose of chemotherapy.
3. Male sex will be excluded.
4. Use of agent designed to suppress ovarian function (i.e. LHRH agonist).
5. Use of exogenous estrogen (hormone replacement therapy) will be prohibited with the exception of topical vaginal preparations (as deemed necessary by the treating physician) and oral contraceptives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Oncology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2005-02; Primary Completion 2009-01-13 (Actual); Study Completion 2009-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Schneider, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States